CLINICAL TRIAL: NCT07034014
Title: A Healthy Volunteer, Single Center, Exploratory Investigation to Evaluate Wearing Properties of Three Different Non-sterile Silicone Self-adhesive Investigational Devices
Brief Title: An Investigation to Evaluate Wearing Properties of Three Different Investigational Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PENGUIN study
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 dressings applied to designated sites on healthy volunteer participants (Other): The investigation will evaluate the dressing and the application regimen.
  Interventions: Device: Dressing

INTERVENTIONS:
Device: Dressing — The dressing will be applied to intact skin on healthy volunteers participants to assess the self-adhesive properties of two investigational devices compared to a test specimen reference. The dressing will be worn for up to 14 days on a designated area on the health volunteers participants back.

SUMMARY:
This clinical investigation will assess the self-adhesive properties of two investigational devices compared to a test specimen reference.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are capable and willing to comply with protocol visits, assessments, and instructions.
* Participants must be in general good health with healthy and intact skin in the test area (as determined by the investigator based on medical history and examination of the application sites).
* Minimal hairiness at the back (location of the application sites).
* Signed written informed consent.

Exclusion Criteria:

* Known allergy/hypersensitivity to the dressing or its components.
* Participants with any features at the application sites will be in contact with the adhesive surface of the dressing, and could influence the investigation.
* Participants not willing to avoid contact of the application sites with water in the morning prior to dressing application and throughout the entire course of the study.
* Participants not willing to avoid applying any detergents to the application sites in the morning prior to dressing application and throughout the entire course of the study.
* Participants not willing to avoid the use of leave on cosmetics such as creams/lotions and sunscreens at the application sites 3 days leading up to dressing application and throughout the entire course of the study.
* Participants not willing to refrain from activities which may directly affect the dressings, application sites or assessments in the morning prior to dressing application and throughout the entire course of the study.
* Participants whose back is not large enough to accommodate all 12 application sites
* Any severe systemic disease that may interfere with the performance, evaluation, and outcome of the investigation as judged by the investigator.
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years.
* Active skin disease at the application sites .
* Any topical medication at the application sites within the last 24 hours prior to the start of the test and/or throughout the entire course of the investigation.
* Pain relief medication on assessment visits . If it is essential for the participant to take pain relief medication on the days mentioned above for any unforeseen reasons, the participant is allowed to use pain relief medication but has to report this to the study center in order to be documented as protocol deviation.
* Pregnancy or lactation.
* Drug addicts, alcoholics.
* AIDS, HIV-positive or infectious hepatitis.
* Individuals who are inmates in psychiatric wards, prison or state institutions, or any individuals otherwise regarded as vulnerable (as per ISO 14155 Section 3.55).
* Participation in another investigative drug or device study currently or within the last 30 days.
* Current participation in a cosmetic study.
* Employees of the investigation sites directly involved in this clinical investigation.
* Employees of the sponsor's company.
* Employees of a competitor company. The participant should not work for any company which produces dressings.
* The participant is considered by the Investigator to be unsuitable to participate in the investigation for any other reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate stay-on-ability of the test specimens compared to the test specimen reference | From enrollment to end of follow-up at day 14.
  The percentage detachment of each test specimen and the test specimen reference will be assessed using a counting grid method. A standardized grid-patterned template will be applied to the application area to objectively quantify the area of detachment. The result will be expressed as a percentage of the total surface area in terms of the mean % detachment at Day 14.
  Unit of Measure: Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Uta Solecke, Principal Investigator — SGS proderm GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Hamburg, Germany